CLINICAL TRIAL: NCT06775860
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study Evaluating the Efficacy and Safety of Oral ICP-332 in Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: ICP-332 in Subjects With Moderate to Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-CL-00604
Record Dates: First submitted 2024-12-25; First posted 2025-01-15 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICP-332 (Experimental)
  Interventions: Drug: ICP-332 Tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: ICP-332 Placebo Tablets

INTERVENTIONS:
Drug: ICP-332 Tablets — ICP-332 will be administered as tablet
  Arms: ICP-332
Drug: ICP-332 Placebo Tablets — ICP-332 Placebo will be administered as tablet
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled phase III study evaluating the efficacy and safety of oral ICP-332 in subjects with moderate to severe atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 75 years of age.
2. Clinical diagnosis of chronic atopic dermatitis (also known as atopic eczema) for at least 1 year
3. Documented recent history of inadequate response to TCS or TCI, or for whom topical treatments are otherwise medically inadvisable.
4. Subjects must meet the following criteria for disease activity:

   * Eczema Area and Severity Index (EASI) score ≥ 16 ;
   * (Body Surface Area )BSA affected by AD ≥ 10% ;
   * (validated Investigator's Global Assessment-AD)vIGA-AD score ≥3 ;
   * Baseline weekly average of daily Worst Pruritus NRS ≥ 4.
5. Women of childbearing potential (WOCBP) and Men must agree

5. Women of childbearing potential (WOCBP) and Men must agree to contraception. 6. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Lack of response or inadequate response to prior treatment with any JAK inhibitor for AD.
2. Other active skin diseases or skin infections requiring systemic treatment or would interfere with appropriate assessment of atopic dermatitis lesions.
3. Pregnant or breastfeeding females.
4. History of any clinically major diseases, with the exception of atopic dermatitis.
5. Consideration by the Investigator, for any reason, that the subject is an unsuitable candidate to receive ICP-332 or participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-11-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving at least a 75% reduction in Eczema Area and Severity Index (EASI 75) from Baseline | 16 weeks
Proportion of subjects achieving Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) of 0 or 1 with at least two grades of reduction from Baseline | 16 weeks

CONTACTS AND LOCATIONS:
Locations (62):
- China (62):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Capital Medical University Affiliated Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Capital Medical University Affiliated Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - The Affiliated Union Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Second Affiliated Hospital of Xiamen Medical College, Xiamen, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Zhongshan University Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - Affiliated Hospital of Hebei University of Engineering, Handan, Hebei
  - Second Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Wuhan Central Hospital, Wuhan, Hubei
  - Wuhan Hospital of Traditional Chinese and Western Medicine (Wuhan No.1 Hospital), Wuhan, Hubei
  - Central South University Xiangya Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Changzhou First People's Hospital, Changzhou, Jiangsu
  - Sir Run Run Hospital, Nanjing Medical University, Nanjing, Jiangsu
  - Yancheng First People's Hospital, Yancheng, Jiangsu
  - The First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Affiliated Hospital of Jiujiang University, Jiujiang, Jiangxi
  - Jiangxi Provincial Dermatology Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shenyang Hospital of Integrated Traditional Chinese and Western Medicine （Shenyang Seventh People's Hospital）, Shenyang, Liaoning
  - Zhongyi Northeast International Hospital Co., Ltd., Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Dermatosis Hospital, Jinan, Shandong
  - Jining First People's Hospital, Jining, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Affiliated Hospital of Tianjin Academy of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Third People's Hospital of Hangzhou, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Fourth Affiliated Hospital, Zhejiang University School of Medicine, Yiwu, Zhejiang